CLINICAL TRIAL: NCT06858735
Title: HYPERION CCA: a Phase 2 Trial of Systemic Therapy With or Without Liver-directed Radiation Therapy for Patients With Advanced Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Varian Medical Systems, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1816; NCI-2025-01520 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Advanced Intrahepatic Cholangiocarcinoma
MeSH Terms: interventions — durvalumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm - Liver-RT + Durvalumab (Experimental): Participants will receive treatment in sequence with standard of care systemic therapy
  Interventions: Drug: Durvalumab
- Standard of Care Arm - Durvalumab + Gemcitabine + Cisplatin (Experimental): Participants will receive treatment in sequence with standard of care systemic therapy
  Interventions: Drug: Durvalumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Durvalumab — Given by IV
Drug: Gemcitabine — Given by IV
  Arms: Standard of Care Arm - Durvalumab + Gemcitabine + Cisplatin
Drug: Cisplatin — Given by IV
  Arms: Standard of Care Arm - Durvalumab + Gemcitabine + Cisplatin

SUMMARY:
This study will compare outcomes for M1 iCCA patients treated with and without L-RT by reviewing iCCA patients found to have M1 disease at initial diagnosis at a single institution between 2010 and 2021 who received L-RT.

DETAILED DESCRIPTION:
Primary Objective:

To assess the overall survival of patients treated with standard of care systemic therapy with or without liver-directed hypofractionated adaptive RT.

Secondary Objectives:

* Patient-reported quality of life as per the FACT-Hep inventory
* Progression-free survival
* Cause of death

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than the age of 18 years old at the time of study entry.
2. Patients with a body mass greater than 30 kg.
3. Patients with a pathological diagnosis of intrahepatic cholangiocarcinoma and at least one intrahepatic tumor measuring 3 cm in greatest dimension
4. Patients must have pathological or radiographic evidence of either:

   c. locally advanced unresectable iCCA - a multidisciplinary discussion should be documented for patients who have liver confined disease, confirming that the patient is not resectable.

   d. extrahepatic metastasis at the time of enrollment - allowable extrahepatic metastases may include disease in non-regional lymph nodes (note that metastatic involvement of regional lymph nodes in the hilum of the liver alone do not qualify as M1 disease), lung, and/or bone.
5. Patients should receive at least 4 cycles of systemic therapy with gemcitabine/cisplatin with durvalumab. If one of the drugs (gemcitabine/cisplatin/durvalumab) was held at any point for medical reasons during the initial 4 cycles, the patient is still eligible as long as the treating team agrees about the ability of the patient to continue systemic therapy.
6. Patients must be appropriate candidates for radiation therapy with adequate liver function, at the discretion of the treating physician.
7. A patient may pre-register at any time before cycle 4 of systemic therapy. To be eligible to pre-register for the trial, they must meet all other inclusion and exclusion criteria, except criteria number 5 regarding the number of cycles of systemic therapy.Pre-registration is not required to enroll.
8. Adequate normal organ and marrow function as defined below:

   Hemoglobin ≥9.0 g/dL Absolute neutrophil count (ANC) ≥1.0 × 109 /L Platelet count ≥75 × 109/L Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.

   AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN

   Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
9. Must have a life expectancy of at least 12 weeks
10. At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at baseline. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to randomization
11. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Participation in another clinical study with an investigational product during the last 1 month.
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
4. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment other than stated in the inclusion criteria. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
5. Major surgical procedure (as defined by the treating physician) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
6. History of allogenic organ transplantation.
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with celiac disease controlled by diet alone
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
9. History of another primary malignancy except for

   1. Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of IP and of low potential risk for recurrence
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated carcinoma in situ without evidence of disease
10. History of leptomeningeal carcinomatosis
11. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry. Patients with brain metastasis or metastases confirmed on imaging will be excluded.
12. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
13. History of active primary immunodeficiency
14. Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of antiHBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Adjust wording as necessary and consider evaluating at screening for studies with known hepatotoxicity or other relevant requirements.

    1. Participants co-infected with HBV and HCV, or co-infected with HBV and HDV, namely: HBV positive (presence of HBsAg and/or anti HBcAb with detectable HBV DNA); AND
    2. HCV positive (presence of anti-HCV antibodies); OR
    3. HDV positive (presence of anti-HDV antibodies). Subjects with HBV infection, characterised by positive HBsAg and/or anti-HBcAb with detectable HBV DNA (≥ 10 IU/ml or above the limit of detection per local laboratory standard), must be treated with antiviral therapy, per institutional practice. Following antiviral therapy initiation, subjects must show adequate viral suppression (ie, HBV DNA ≤ 2000 IU/mL) as prior to randomisation. Participants will remain on antiviral therapy for the study duration and for 6 months after the last dose of IP.
    4. Subjects with HBV infection, characterised by positive HBsAg and/or anti-HBcAb with undetectable HBV DNA (< 10 IU/ml or under the limit of detection per local lab standard) do not require antiviral therapy prior to randomisation. These subjects will be tested at every cycle to monitor HBV DNA levels; if HBV DNA is detected (≥ 10 IU/ml or above the limit of detection per local lab standard), antiviral therapy must be initiated, continued for the study duration and for 6 months after the last dose of IP.
15. Known HIV infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA load for 6 months, CD4+ count of >200, no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 6 months on the same anti HIV medications.
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90days after the last dose of IP.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
21. Patients who have received prior anti-PD-1 or anti PD-L1:

    1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    3. Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
22. Judgment by the treating physician that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-11-19 (Estimated); Study Completion 2030-11-19 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Koay, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org